CLINICAL TRIAL: NCT04729322
Title: Pilot Trial of Fecal Microbiota Transplantation and Re-Introduction of Anti-PD-1 Therapy in dMMR Colorectal Adenocarcinoma Anti-PD-1 Non-Responders
Brief Title: Fecal Microbiota Transplant and Re-introduction of Anti-PD-1 Therapy (Pembrolizumab or Nivolumab) for the Treatment of Metastatic Colorectal Cancer in Anti-PD-1 Non-responders
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2020-0186; NCI-2020-13897 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2020-0186 (Other: M D Anderson Cancer Center); P50CA221707 (NIH)
Record Dates: First submitted 2021-01-08; First posted 2021-01-28 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Metastatic Colorectal Adenocarcinoma; Metastatic Small Intestinal Adenocarcinoma; Stage IV Colorectal Cancer AJCC v8; Stage IV Small Intestinal Adenocarcinoma AJCC v8; Stage IVA Colorectal Cancer AJCC v8; Stage IVB Colorectal Cancer AJCC v8; Stage IVC Colorectal Cancer AJCC v8
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Biopsy; Fecal Microbiota Transplantation; Parturition; Metronidazole; Benchmarking; Neomycin; Nivolumab; pembrolizumab; Vancomycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm I (FMT, pembrolizumab) (Experimental): Patients receive metronidazole PO Q8H on days -14 to -8 and then vancomycin PO Q6H and neomycin PO Q6H on days -8 to -6. Patients then undergo colonoscopic FMT on day -5.
  POST-COLONOSCOPIC FMT: Patients receive standard of care pembrolizumab IV over 30 minutes on day 1. Patients also receive fecal microbiota transplantation capsule PO on days 1, 8, and 15 of cycle 1. Beginning in cycle 2, patients receive fecal microbiota transplantation capsule PO on day 1. Cycles repeat every 21 days for up to 6 months in the absence of disease progression or unacceptable toxicity.
  Interventions: Procedure: Biopsy; Procedure: Fecal Microbiota Transplantation; Drug: Fecal Microbiota Transplantation Capsule; Drug: Metronidazole; Drug: Neomycin; Biological: Pembrolizumab; Other: Questionnaire Administration; Drug: Vancomycin
- Arm II (FMT, nivolumab) (Experimental): Patients receive metronidazole PO Q8H on days -14 to -8 and then vancomycin PO Q6H and neomycin PO Q6H on days -8 to -6. Patients then undergo colonoscopic FMT on day -5.
  POST-COLONOSCOPIC FMT: Patients receive standard of care nivolumab IV over 30 minutes on day 1. Patients also receive fecal microbiota transplantation capsule PO on days 1 and 8 of cycles 1-2. Beginning in cycle 4, patients receive fecal microbiota transplantation capsule PO on day 1 of every other cycle. Cycles repeat every 14 days for up to 6 months in the absence of disease progression or unacceptable toxicity.
  Interventions: Procedure: Biopsy; Procedure: Fecal Microbiota Transplantation; Drug: Fecal Microbiota Transplantation Capsule; Drug: Metronidazole; Biological: Nivolumab; Other: Questionnaire Administration; Drug: Vancomycin

INTERVENTIONS:
Procedure: Biopsy — Undergo biopsy
  Other Names: BIOPSY_TYPE; Bx
Procedure: Fecal Microbiota Transplantation — Undergo colonoscopic FMT
  Other Names: Fecal Material Transplantation; Fecal Transplantation; FMT; Poo Transplant; Poop Transplant; Stool Transplant
Drug: Fecal Microbiota Transplantation Capsule — Given PO
  Other Names: Fecal Microbiota Preparation Delivery Capsule; FMPCapDE; FMT Capsule DE; FMT Capsule Delivery; FMT DE Capsule
Drug: Metronidazole — Given PO
  Other Names: Flagyl; Flagyl I.V. RTU; Tricom
Drug: Neomycin — Given PO
  Other Names: Neomycin Complex
  Arms: Arm I (FMT, pembrolizumab)
Biological: Nivolumab — Given IV
  Other Names: BMS-936558; MDX-1106; NIVO; ONO-4538; Opdivo
  Arms: Arm II (FMT, nivolumab)
Biological: Pembrolizumab — Given IV
  Other Names: Keytruda; Lambrolizumab; MK-3475; SCH 900475
  Arms: Arm I (FMT, pembrolizumab)
Other: Questionnaire Administration — Ancillary studies
Drug: Vancomycin — Given PO

SUMMARY:
This phase II trial studies the effect of fecal microbiota transplant and re-introduction of anti-PD-1 therapy (pembrolizumab or nivolumab) in treating anti-PD-1 non-responders with colorectal cancer that has spread to other places in the body (metastatic). Fecal microbiota transplants contain the normal bacteria and viruses found in fecal (stool) material. Immunotherapy with monoclonal antibodies, such as pembrolizumab and nivolumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. Giving pembrolizumab or nivolumab with fecal microbiota transplants may help to control the disease.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To evaluate the efficacy of pembrolizumab or nivolumab in conjunction with fecal microbiota transplant (FMT) from PD-1 responding mismatch-repair deficiency (dMMR) colorectal cancer (CRC) patients for treatment of PD-1 non-responding dMMR CRC patient.

ELIGIBILITY:
Eligibility Criteria:

Participant Inclusion Criteria:

Participants are eligible to be included in the study only if all of the following criteria apply:

1. At least 18 years of age on the day of signing informed consent
2. Histologically/cytologically confirmed diagnosis of solid tumor
3. Tumor that is deficient in mismatch repair (dMMR) or microsatellite instability high (MSI-H) as determined by one of three methods:

   1. Immunohistochemistry determined dMMR by complete loss of MLH1, PMS2, MSH2 or MSH6
   2. PCR determined microsatellite instability at >30% of tested microsatellites
   3. Next-generation determined MSI-H based upon instability at multiple microsatellites as determined by the specific next generation sequencing panel
4. Have metastatic disease that is measurable based on iRECIST v1.1.
5. Demonstrated prior progression on anti-PD1/L1 based therapy by radiographic progression. The potential for psuedoprogression should be excluded by concurrent carcinoembryonic antigen (CEA) or other tumor marker or ctDNA elevation, or clinical symptom progression, or short interval repeat imaging confirming progression.

   1. Must have received at least 2 doses of a PD1/PD-L1 inhibitor
   2. Progressive disease either during therapy or within 2 months of last dose of therapy.
6. An Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1.
7. Patients must be willing to undergone mandatory tumor biopsies at pre-treatment, at time of colonoscopy if possible and on-treatment (unless deemed unsafe by interventional radiology or by approval by study PI).
8. The participant (or legally acceptable representative if applicable) provides written informed consent for the trial.
9. Estimated life-expectancy of > 4 months.
10. Adequate hematological function, defined by white blood cell (WBC) count ≥ 3,000/microL, platelet count ≥75,000/microL, and Hgb ≥ 8 g/dL.
11. Adequate hepatic function defined by a total bilirubin level ≤ 1.5 × the upper limit of normal (ULN)[except if Gilberts syndrome and then total bilirubin ≤ 3x is allowed], an AST, level ≤ 2.5 × ULN, and an ALT level ≤ 2.5 × ULN. If liver metastases are present, then AST and ALT levels must be ≤ 4 × ULN
12. Adequate renal function defined by an estimated creatinine clearance >30 mL/min according to the Cockcroft-Gault formula or by a creatinine clearance measurement from a 24-hour urine collection.
13. Highly effective contraception for both male and female subjects if the risk of conception exists. Highly effective contraception must be used 30 days prior to first study-drug administration, for the duration of trial treatment, and for at least for 6 months (women and men after taking your last dose of any of the trial drugs (see Appendix 3 for further details). Should a female patient (or male patient's sexual partner) become pregnant or should either the female patient (or male patient's partner) suspect she is pregnant while the patient's study-participation is ongoing, the treating physician should be informed immediately.

Participant Exclusion Criteria:

Participants are excluded from the study if any of the following criteria apply:

1. Has received prior systemic anti-cancer therapy including investigational agents within 2 weeks of study treatment (excluding continuation of ongoing nivolumab or pembrolizumab therapy).
2. If participant received major surgery within last 4 weeks, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting study treatment.
3. Has an ileostomy or colostomy bag.
4. Has received prior radiotherapy within 2 weeks of start of study treatment. Participants must have recovered from all radiation-related toxicities (excluding skin toxicity), not require corticosteroids, and not have had radiation pneumonitis.
5. Has received a live vaccine within 30 days prior to the first dose of study drug. Examples of live vaccines include, but are not limited to, the following: measles, mumps, rubella, varicella/zoster (chicken pox), yellow fever, rabies, Bacillus Calmette-Guérin (BCG), and typhoid vaccine. Seasonal influenza vaccines for injection are generally killed virus vaccines and are allowed; however, intranasal influenza vaccines (e.g., FluMist®) are live attenuated vaccines and are not allowed.
6. Has a diagnosis of immunodeficiency (excluding IgA deficiency).
7. Has an active autoimmune condition and is receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior to the first dose of study drug.

   1. Subjects requiring hormone replacement with corticosteroids are eligible if the steroids are administered only for the purpose of hormonal replacement and at doses ≤ 10mg of prednisone or equivalent per day.
   2. Administration of steroids for other conditions through a route known to result in a minimal systemic exposure (topical, intranasal, intro-ocular, or inhalation) is acceptable.
8. Has severe hypersensitivity (≥Grade 3) to pembrolizumab or nivolumab and/or any of its excipients.
9. Serious adverse immune related adverse events (grade 3 or 4) with previous immune checkpoint therapy, that were symptomatic and required prolong immunosuppression (>6weeks).
10. Has an active infection requiring systemic therapy.
11. Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the subject's participation for the full duration of the study, or is not in the study subject's best interest to participate, in the opinion of the treating investigator.
12. Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
13. Pregnant or nursing women
14. For women of childbearing age, a positive urine pregnancy test within 72 hours prior to enrollment. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2021-02-22 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Objective response rate | Up to 3 years post-treatment
  Assessed by Immune-Modified Response Evaluation Criteria in Solid Tumors (iRECIST). Will be summarized by mean, standard error, and 95% confidence interval.

CONTACTS AND LOCATIONS:
Overall Officials: Michael J Overman, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: M D Anderson Cancer Center — http://www.mdanderson.org

DOCUMENTS (1):
  • Informed Consent Form (2023-05-01): https://cdn.clinicaltrials.gov/large-docs/22/NCT04729322/ICF_000.pdf